CLINICAL TRIAL: NCT03279718
Title: Exploring Efficacy of Periodontal Treatment on Systemic Inflammation and for Prevention of Exacerbations in Patients With Chronic Obstructive Pulmonary Disease (COPD): A Pilot Study
Brief Title: Efficacy of Periodontal Treatment on Systemic Inflammation and for Prevention of Exacerbations in Patients With COPD
Acronym: Expertention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges due to COVID pandemic
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Michael Kreuter, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Expertention
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: COPD Exacerbation, Periodontal Health
MeSH Terms: interventions — Periodontal Index

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periodontal treatment (Experimental)
  Interventions: Procedure: Periodontal Treatment
- only oral hygiene instruction, no treatment (No Intervention)

INTERVENTIONS:
Procedure: Periodontal Treatment — Scaling and root planing
  Arms: periodontal treatment

SUMMARY:
Current data are showing a potential link between inflammatory biomarkers in chronic periodontitis and COPD. However the impact of periodontal treatment on systemic inflammation as measured by biomarkers and time to occurrence of acute exacerbations (AECOPD) remains an important but unresolved issue. This pilot study will provide information on effects of periodontal treatment on systemic inflammation and the course of COPD including acute exacerbation.

40 patients with chronic periodontitis and COPD will be included in this study. First baseline information (age, gender, lifestyle, smoking history, medical history, medication, frequency of exacerbation, dental treatments) are recorded. Then patient's health status is assessed using the COPD Assessment Test (CAT) and a comprehensive lung function testing (bodyplethysmograph) is conducted to assess lung functional severity of COPD. Blood samples are taken for analysis of various inflammatory biomarkers and saliva and sputum samples are collected for analysis of microbiome.

Afterwards experienced dentists will conduct oral health examination and record the periodontal conditions of every patient. Samples of gingival crevicular fluid for determining Matrix metallopeptidase 8 (MMP8), Interleukin 1 beta (IL-1beta) and Interleukin 6 (IL-69 levels and for microbiome analysis will be taken. After randomization to one of the two study groups (intervention group: periodontal treatment / control group: no periodontal treatment) all patients get comprehensive oral hygiene instructions, irrespective of their periodontal status . Patients of the control group receive no further planned dental intervention. For patients of the experimental group, who need periodontal treatment due to the presence of periodontal pocket depth of ≥ 4 mm an appropriate care plan will be determined and supra- and subgingival scaling and root planing will be performed.

During a 3, 6 and 12 months follow-up patient's current health condition will be assessed using the CAT. Additionally lung function tests (bodyplethysmograph) will be performed and clinical periodontal parameters are re-evaluated. To detect and assess COPD exacerbations in this trial, patients will complete a daily diary during the whole follow-up period which will be provided to the clinical researcher at each study visit. Furthermore the cough and sputum assessment questionnaire (CASA-Q)) will be used at each telephone call and at each visit in the pulmonary center. After 6 and 12 months blood, sputum, saliva and gingival crevicular fluid will be taken additionally. To understand the microbial ecology mechanisms linking periodontitis to COPD combined analysis of oral cavity microbiome (GCF) and lung microbiome (sputum) will be conducted. The biomarkers high sensitive C-reactive Protein (hsCRP), MMP8, IL-1beta und IL-6 will be determined in blood and in gingival crevicular fluid, respectively.

ELIGIBILITY:
Inclusion Criteria:

COPD functional class B to D (moderate to very severe) according to the Global Initiative For Chronic Obstructive Lung Disease (GOLD)

* age ≥ 40 and ≤ 80 years
* at least 10 natural teeth
* COPD-associated hsCRP elevation (after exclusion of infection) with hsCRP > 3mg/l
* presence of chronic periodontitis
* at least 1 exacerbation leading to treatment with systemic glucocorticoids or antibiotics or hospitalization within the last 12 months
* non-smoker or ex-smoker for at least the last 6 months
* ability to understand the character and individual consequences of participation in this trial and to give written informed consent
* provision of a written informed consent to participation in the trial prior to trial start and any trial-related procedures

Exclusion Criteria:

* any subgingival root-planing or any kind of periodontal surgery within the last 6 months (professional tooth cleaning is allowed)
* any antibiotics and/or systemic corticosteroid medication in the last 4 weeks before inclusion
* any antibiotics needed as prophylaxis or as an adjunct to periodontal treatment
* diagnostical bronchoscopy within the last 8 weeks
* any kind of bronchoscopy and lung surgery (volume reduction, transplantation, pneumonectomy) within the last 6 months
* concurrent participation in any interventional clinical trial (observational trials are allowed)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in blood serum inflammatory biomarker hsCRP | after 6 months and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kreuter, Prof., Principal Investigator — Thoraxklinik, University Hospital Heidelberg
Locations (3):
- Germany (3):
  - Clinic for Operative Dentistry, University Hospital Heidelberg, Heidelberg
  - Medical Center for Dental and Oral Medicine, Dept. of Periodontology, Philipps-University of Marburg, Marburg
  - Clinic for Internal Medicine (focus Pneumology) , University Hospital Gießen und Marburg, Marburg